CLINICAL TRIAL: NCT06676254
Title: Role of HbA1c in Predicting Adverse Pregnancy Outcomes Among Gestational Diabetes Mellitus Women: a Retrospective Study
Brief Title: Role of HbA1c in Predicting Adverse Pregnancy Outcomes
Status: Recruiting | Type: Observational
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Rahana Abd Rahman, Assoc Prof Dr, National University of Malaysia
Other Study IDs: JEP-2024-475
Record Dates: First submitted 2024-08-12; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Gestational Diabetes
Keywords: HbA1c; Gestational diabetes; large for gestational age; shoulder dystocia; caesarean section
MeSH Terms: conditions — Diabetes, Gestational; Shoulder Dystocia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum levels of HbA1c and fructosamine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the reference value of HbA1c that can be used to predict adverse pregnancy outcomes. These adverse outcomes include LGA fetus, shoulder dystocia, caesarean section, pre-term birth, pre-eclampsia and fetal neonatal hypoglycaemia.

DETAILED DESCRIPTION:
This study involves the data in our centre concerning women with gestational diabetes mellitus. The diagnosis of gestational diabetes mellitus is based on NICE guideline whereby the fasting glucose is 5.6 mol/l or more and 2 hours post glucose load 7.8 mol/l or more. The results of HbA1c and fructosamine taken during the antenatal care are documented. Outcomes of the pregnancy are documented such as antenatal complications, mode of delivery, gestational age at delivery, intrapartum and postpartum complications and neonatal complications. The results of this study is hoped to provide information on the optimum targeted levels of HbA1c and fructosamine for patients with gestational diabetes mellitus. This is the gap in knowledge in managing this cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman with singleton pregnancy
* Confirmed diagnosis of GDM based on Malaysia CPG (≥5.1/7.8)
* HbA1c level taken at least once at any time during the pregnancy
* Delivery after 28 weeks gestation

Exclusion Criteria:

* Major fetal anomaly
* Haemoglobin level of ≤9 g/dL (moderate or severe anaemia in pregnancy)
* Women with autoimmune diseases
* Overt diabetes or pre-existing diabetes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Antenatal women attended antenatal clinics between January 2020-June 2024 in Hospital Canselor Tuanku Muhriz and diagnosed with GDM will be included in the study using purposive sampling method. Diagnosis of GDM is based on the Malaysia Diabetes CPG Guideline (fasting plasma glucose ≥5.1, 2 hours post-prandial ≥7.8).
Sampling Method: Non-Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
To determine the HbA1c reference value in predicting adverse pregnancy outcomes | Throughout study up to 1 year
  c) To determine the HbA1c value to be used at each trimester in predicting adverse pregnancy outcomes

SECONDARY OUTCOMES:
To determine the prevalence of adverse pregnancy outcomes among women with GDM | Throughout study up to 1 year
  Measurement of prevalent
To assess the HbA1c value during the diagnosis of GDM and its association with adverse pregnancy outcomes | Throughout study up to 1 year
  Relationship between HbA1c and adverse pregnancy outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics & Gynaecology, Hospital Canselor Tuanku Muhriz, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No